CLINICAL TRIAL: NCT05706818
Title: Validity and Reliability of the Turkish Version of the Community Integration Questionnaire-Revised (CIQ-R) in Lower Limb Amputees
Brief Title: Validity and Reliability of the Community Integration Questionnaire-Revised in Lower Limb Amputees
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Serdar Y ESEN, Pirincipal investigator, Hacettepe University
Other Study IDs: GO 19/1039
Record Dates: First submitted 2023-01-18; First posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Amputation
Keywords: lower limb amputees; community integration; social participation; validity; reliability

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Validity and reliability study — Validity and reliability assessment of the Community Integration Questionnaire-revised

SUMMARY:
The goal of this clinical trial is to determine the validity and reliability of the Community Integration Questionnaire-Revised (CIQ-R) scale in lower limb amputees. The main questions it aims to answer are:

* The Turkish version of the Community Integration Questionnaire-Revised is valid for lower extremity amputees.
* The Turkish version of the Community Integration Questionnaire-Revised is reliable for lower extremity amputees.

Participants will:

• Fill out general information, CIQ-R, TAPES, and ABIS forms.

DETAILED DESCRIPTION:
The aim of this study is to determine the validity and reliability of the Community Integration Questionnaire-Revised (CIQ-R) scale in lower limb amputees. Lower limb amputees aged 18-65 years who used prostheses for at least 6 months and volunteered to participate in the study were included in the study. The adaptation of amputees to prostheses was evaluated with the "Trinity Amputation and Prosthesis Experience Scale" (TAPES), their perception of physical appearance with the "Amputee Body Image Scale" (ABIS), and their community integration with the CIQ-R. Correlation with TAPES and ABIS and confirmatory factor analysis were performed to determine the construct validity of the CIQ-R scale. The test-retest reliability of the CIQ-R scale was determined by the intraclass correlation coefficient (ICC) method. Internal consistency analysis was evaluated with Cronbach's alpha. 90 amputees were included in the study (mean age: 40.96±12.89 years; BMI: 25.55±5.5 kg/m2). The CIQ-R scale was reapplied to 18 of the participants 1 week later.

ELIGIBILITY:
Inclusion Criteria:

* Those between the ages of 18 and 65
* Lower extremity amputation
* Use of a prosthesis for at least one year
* Individuals who volunteered to participate in the research.

Exclusion Criteria:

* Have any known cognitive problems
* Illiterate individuals were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lower extremity amputees between the ages of 18 and 65 with a prosthesis usage period of more than 1 year who can speak and read Turkish.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2022-03-27 (Actual)

PRIMARY OUTCOMES:
The Community Integration Questionnaire-Revised | 1st day
  The Community Integration Questionnaire-Revised (CIQ-R) is a self-report, standardized instrument designed to assess an individual's degree of community integration. On this multisectional scale, patients get a minimum of 0 points (worst condition) and a maximum of 35 points (best condition).
The Community Integration Questionnaire-Revised | 5 days later
  The Community Integration Questionnaire-Revised (CIQ-R) is a self-report, standardized instrument designed to assess an individual's degree of community integration. On this multisectional scale, patients get a minimum of 0 points (worst condition) and a maximum of 35 points (best condition).
Trinity Amputation and Prosthesis Experience Scales | 1st day
  The Trinity Amputation and Prosthesis Experience Scales (TAPES) is a self-administered questionnaire that comprises psychosocial adjustment, activity restriction, and prosthetic satisfaction domains, each with three subscales.
The Amputee Body Image Scale | 1st day
  The Amputee Body Image Scale affects the individual's perception of their own physical condition, life satisfaction, and well-being. The ABIS consists of 20 items and is scored on a 5-point Likert scale. Three items (3, 12, and 16) are reverse scored. The total score varies between 20-100. A high score indicates poor body image.

CONTACTS AND LOCATIONS:
Overall Officials: Serdar Y ESEN, MSc, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Callaway L, Winkler D, Tippett A, Herd N, Migliorini C, Willer B. The Community Integration Questionnaire - Revised: Australian normative data and measurement of electronic social networking. Aust Occup Ther J. 2016 Jun;63(3):143-53. doi: 10.1111/1440-1630.12284. Epub 2016 Apr 13. PMID 27072343
- [Background] Topuz S, Ulger O, Yakut Y, Gul Sener F. Reliability and construct validity of the Turkish version of the Trinity Amputation and Prosthetic Experience Scales (TAPES) in lower limb amputees. Prosthet Orthot Int. 2011 Jun;35(2):201-6. doi: 10.1177/0309364611407678. PMID 21697202
- [Background] Bumin G, Bayramlar K, Yakut Y, Sener GY. Cross cultural adaptation and reliability of the Turkish version of Amputee Body Image Scale (ABIS). J Back Musculoskelet Rehabil. 2009;22(1):11-6. doi: 10.3233/BMR-2009-0208. PMID 20023358